CLINICAL TRIAL: NCT07368088
Title: A Clinical Study of Advanced Regenerative Medicine to Evaluate the Safety and Potential Efficacy of PNEUMOSTEM® for Improving Respiratory Outcomes in Very Premature Infants Diagnosed With Early Pulmonary Arterial Hypertension
Brief Title: PNEUMOSTEM® for Improving Respiratory Outcomes in Very Premature Infants Diagnosed With Early Pulmonary Arterial Hypertension
Acronym: REVIVE-PH
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, So Yoon Ahn, Clinical Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-10-080
Record Dates: First submitted 2025-11-25; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Arterial Hypertension (PAH); Premature Infants
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Premature Birth

STUDY DESIGN:
Intervention Model Description: Single center, Single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PNEUMOSTEM® treatment arm (Experimental): PNEUMOSTEM® will be administered intratracheally as a single dose of 2.0x10,000,000 cells/kg on Day 1.
  Interventions: Biological: PNEUMOSTEM®

INTERVENTIONS:
Biological: PNEUMOSTEM® — PNEUMOSTEM® will be administered intratracheally as a single dose of 2.0x10000000 cells/kg on Day 1.
  Other Names: Cell therapy product

SUMMARY:
The goal of this clinical trial is to evaluate the safety and potential efficacy of PNEUMOSTEM® for improving respiratory outcomes in very premature infants diagnosed with Early Pulmonary Arterial Hypertension. The main questions it aims to answer are:

* In very premature infants diagnosed with early pulmonary arterial hypertension, will a single intratracheal administration of PNEUMOSTEM®(Allogeneic umbilical cord blood-derived mesenchymal stem cells) result in improvement of pulmonary arterial hypertension based on echocardiographic assessment?
* In very premature infants diagnosed with early pulmonary arterial hypertension who show improvement of pulmonary arterial hypertension based on echocardiographic assessment following a single intratracheal administration of PNEUMOSTEM®(Allogeneic umbilical cord blood-derived mesenchymal stem cells), at what time point does this improvement occur?

Participants will:

* Single intratracheal dose of PNEUMOSTEM® at 2.0 x 10,000,000 cells/kg
* Acute adverse event monitoring: 24 hours post-administration for safety assessment
* Follow- up time points: Day 1(Baseline, PNEUMOSTEM® administration), Day 2, Week 1, Week 2, Postnatal Day 28, PMA 36~40 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Premature infants within 2 weeks of birth with a gestational age of 28 weeks or less or birth weight of less than 1,250g who require continuous invasive mechanical ventilation
2. When diagnosed with early pulmonary arterial hypertension satisfying condition ① or ② up to 14 days after birth:

   * When on or more of the following abnormal findings are present on echocardiography performed between 4 and 14 days after birth (findings at 1-3 days after birth correspond to early neonatal transition):

     1. Sytemic or suprasystemic pulmonary artery pressure >40mmHg(based on peak Doppler velocity of tricuspid regurgitation)
     2. Right-to-left or bidirectional shunt through patent ductus arteriosus, foramen ovale, or atrial septal defect
     3. Flattened interventricular septum or D-shaped left ventricle at end systole ② When receiving nitric oxide(NO) inhalation therapy for persistent pulmonary hypertension of the newborn(PPHN) within 3 days after birth

Exclusion Criteria:

1. Those witth cyanotic congenital heart defects or acyanotic congenital heart defects causing heart failure, excluding patent ductus arteriosus in premature infatns
2. Those with severe pulmonary malformations such as congenital diaphragmatic hernia or congenital cystic lung disease
3. Those who underwent surgery within 72 hours before or after administration of the investigational cell product, or those for whom surgery is anticipated
4. Those who received surfactant within 24 hours prior to administration of the investigattional cell product
5. Those with chromosomal abnormalities accompanied by severe malformations(such as Edwards syndrome, Patau syndrome, Down syndrome, etc.) and severe congenital malformations(such as hydrocephalus, encephalocele, etc.)
6. Those with severe congenital infectious diseases(such as herpes, toxoplasmosis, rubella, syphilis, AIDS, etc.)
7. Those with severe sepsis or shock due to active infection not adequately treated with antibiotics
8. Those who have a history of participation in other advanced regenerative medicine clinical studies or clinical trials
9. Others deemed inappropriate by tthe investigator to participate in this advanced regenerative medicine clinical study

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Time point(week) of complete reversal of cardiac shunt direction | Biweekly from day after PNEUMOSTEM administration until postnatal day 28
  Time from PNEUMOSTEM administration to complete reversal of intracardiac shunt from right-to-left to complete left-to-right direction, as assessed by echocardiography.
Time to normalization of ventricular septal configuration | Once between postnatal day 28 and PMA 36~40 weeks
  Time from PNEUMOSTEM administration to resolution of flattened interventricular septum or disappearance of D-shaped left ventricle at end-systole, as assessed by echocardiography.
Change in duration of pulmonary hypertension medication use | Daily on PNEUMOSTEM administration day and the next day
  Change in duration of pulmonary hypertension medication use by medication type following PNEUMOSTEM administration compared to standard care. Duration will be measured in days for each medication type used to treat pulmonary hypertension.
Change in duration of mechanical ventilation | Weekly at week 1 and week 2 after PNEUMOSTEM administration
  Change in total duration of mechalical ventilator use following PNEUMOSTEM andministration compared to standard care. Duration will be measured in days from initiation to discontinuation of mechanical ventilation.
Change in duration of supplemental oxygen therapy. | Weekly at week 1 and week 2 after PNEUMOSTEM administration
  Change in total duration of supplemental oxygen use following PNEUMOSTEM administration compared to standard care. Duration will be measured in days from initiation to discontinuation of oxygen therapy.
Incidence of Bronchopulmonary Dysplasia(BPD) | At postnatal day 28 and at between PMA 36~40 weeks
  Inicidence of bronchopulmonary dysplasia assessed according to standard diagnostic criteria(requirement for supplemental oxygen at 28 days of postnatal age and/or at 36 weeks postmenstrual age).
Severity of Bronchopulmonary Dysplasia(BPD) | At postnatal day 28 and at between PMA 36~40 weeks
  Severity assessment of bronchopulmonary dysplasia categorized according to the definition of NIHCD 2001, NICHD 2018 and JENSEN 2019.
Incidence of Retinopathy of Prematurity(ROP) | Once at between PMA 36~40 weeks
  Incidence of retinopathy of prematurity assessed by ophthalmologic examination according to the International Classification of Retinopathy of Prematurity.
Severity of Retinopathy of Prematurity(ROP) | Once at between PMA 36~40 weeks
  Severity assessment of retinopathy of prematurity including staging(Stage 1~5), zone(Zone I, II, or III), and presence of pulse disease. Assessment of treatment requirements including lase photocoagulation, anti-VEGF injection, or surgical intervention.
Time point of brain injury ditection on Brain MRI | Once at between PMA 36~40 weeks
  Time point of early detection of brain injury or neurodevelopmental abnormalities on brain MRI performed at postmenstrual age 36~40 weeks. Brain injuries assessed include intraventricular hemorrhage, periventricular leukomalacia, and other structural abnormalities.
Incidence of Respiratory-related mortality | From PNEUMOSTEM administration to PMA 36~40 weeks
  Incidence of respiratory-related moratlity confirmed by medical records and information survey. Respiratory-related mortality is defined as death primarily attributed to respiratory failure, pulmonary hypertension, or complications of bronchopulmonary dysplasia.
Tiem point of respiratory-related mortality | From PNEUMOSTEM administration to PMA 36~40 weeks
  Postnatal age(in days) at which respiratory-related death occurs in participants who experience this outcome. Time will be measured from PNEUMOSTEM administration to the date of death.

SECONDARY OUTCOMES:
Incidence of Adverse Events Assessed by latest version of CTCAE | From PNEUMOSTEM administration to PMA 36~40 weeks
  Incidence of adverse events graded according to the latest version of Common Terminology Criteria for Adverse Events(CTCAE). All adverse events will be recorded and categorized by system organ class and severity grade.
Change in anthropometric measurements - Weight | From PNEUMOSTEM administration to PMA 36~40 weeks
  Change in body weight from baseline(PNEUMOSTEM administration day) measured in grams.
Change in anthropometric measurements - Head Circumference | From PNEUMOSTEM administration to PMA 36~40 weeks
  Change in head circumference from baseline(PNEUMOSTEM administration day) measured in centimeters.
Abnormal findings on physical examination - Skin and Head/Neck | From PNEUMOSTEM administration to PMA 36~40 weeks
  Incidence of clinically significant abnormal findings on physical examination of skin and head/neck regions.
Abnormal findings on physical examination - Cardiovascular and Respiratory systems | From PNEUMOSTEM administration to PMA 36~40 weeks
  Incidence of clinically significant abnormal findings on physical examination of heart and lung systems.
Abnormal findings on physical examination - Abdomen and Genitalia | From PNEUMOSTEM administration to PMA 36~40 weeks
  Incidence of clinically significant abnormal findings on physical examination of abdomen and genitalia.
Abnormal findings on physical examination - Nervous and Musculoskeletal systems | From PNEUMOSTEM administration to PMA 36~40 weeks
  Incidence of clinically significant abnormal findings on physical examination of nervous system and musculoskeletal systems.
Change in vital signs - Blood pressure | From PNEUMOSTEM administration to PMA 36~40 weeks
  Change in systolic and diastolic blood pressure from baseline(PNEUMOSTEM administration day) measured in mmHg.
Change in vital signs - Body temperature | From PNEUMOSTEM administration to PMA 36~40 weeks
  Change in body temperature from baseline(PNEUMOSTEM administration day) measured in degrees celsius.
Change in vital signs - Heart rate | From PNEUMOSTEM administration to PMA 36~40 weeks
  Change in heart rate(pulse) from baseline(PNEUMOSTEM administration day) measured in beats per minute.
Change in vital signs - Respiratory rate | From PNEUMOSTEM administration to PMA 36~40 weeks
  Change in respiratory rate from baseline(PNEUMOSTEM administration day) measured in breaths per minute.
Change in vital signs - Oxygen saturation | From PNEUMOSTEM administration to PMA 36~40 weeks
  Change in oxygen saturation(SpO2) from baseline(PNEUMOSTEM administration day) measure as percentage.
Abnormal laboratory values - Hematology | Once at screening
  Incidence of clinically significant abnormal hematology laboratory values including white blood cell count(WBC), red blood cell count(RBC), hemoglobin(Hb), hematocrit(Hct), and platelet count(PLT).
Abnormal laboratory values - Blood chemistry | At screening and within 24 hours after PNEUMOSTEM administration
  Incidence of clinically significant abnormal blood chemistry values including C-reactive protein(CRP) and other relevant biochemical markers.
Abnormal Electrocardiography findings | From PNEUMOSTEM administration to PMA 36~40 weeks
  Incidence of clinically significant abnormal findings on continuous electrocardiography monitoring including arrhythmias, conduction abnormalities, or other cardiac electrical disturbances.
Incidence of infectious disease | At screening and weekly from baseline(PNEUMOSTEM adminitration day) to week 2
  Incidence of infectious disease identified by blood and tracheal aspirate(TTA) cultures with component analysis and pathogen identification.
Abnormal blood gas analysis | From PNEUMOSTEM administration to postnatal day 28
  Incidence of clinically significant abnormal blood gas analysis results for assessment of respiratory and metabolic status including PH, PaO2, PaCO2 and base excess.
Abnormal findings on chest x-ray | At screening, within 24 hours after PNEUMOSTEM adminitration, a week after PNEUMOSTEM administration, postnatal day 28 and at between PMA 36~40 weeks
  Incidence of clinically significant abnormal findings on chest radiography including evaluation for pleural effusion, pneumothorax, infiltrates, or other pulmonary abnormalities.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, 81, Irwon-ro, Gangnam-gu, Seoul, Republic of Korea, Seoul, South Korea